CLINICAL TRIAL: NCT07312526
Title: Shanghai Clinical Cohort - Esophageal Cancer Cohort
Brief Title: Shanghai Clinical Cohort - Esophageal Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Collaborators: Shanghai Zhongshan Hospital (Other); Shanghai Cancer Hospital, China (Other); Changhai hospital of Navy Medical University (Unknown)
Responsible Party: Principal Investigator, Zhigang Li, Prof., Shanghai Chest Hospital
Other Study IDs: IS25163
Record Dates: First submitted 2025-11-17; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Esophageal Cancer; Esophagectomy
Keywords: esophageal cancer; esophagecomy
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Esophagectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: esophagectomy — esophagectomy

SUMMARY:
A prospective cohort of patients who received esophagectomy for esophageal cancer in participating centers.

DETAILED DESCRIPTION:
A prospective cohort of patients who received esophagectomy for esophageal cancer in participating centers.

ELIGIBILITY:
Inclusion Criteria:

* Received esophagectomy in these centers for esophageal cancer.

Exclusion Criteria:

* No esophagectomy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients received esophagectomy for esophageal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 2116 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overal survival | From the date of enrollment until the date of death or loss of follow-up, assessed up to 10 years. Follow-up is scheduled every 3 months in the first 2 years. Every 6 months from the 2nd to the 5th year. Then once a year. Until death or loss of follow.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No